CLINICAL TRIAL: NCT05675930
Title: A Multi-Center, Phase II, Randomized Double-Blind Trial to Evaluate the Efficacy and Safety of Photobiomodulation for the Treatment of Oral Chronic Graft-Versus-Host Disease After Allogeneic Stem Cell Transplantation (the LIGHT Trial)
Brief Title: A Study of Photobiomodulation (PBM) Therapy in People With Oral Graft-Versus-Host Disease (GVHD) After Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-271
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Graft-Versus-Host Disease; GVHD; Undefined
Keywords: Graft-Versus-Host Disease; GVHD; Chronic Graft Versus Host Disease Oral; PhotobiomoduLatIon; Memorial Sloan Kettering Cancer Center; 22-271
MeSH Terms: conditions — Graft vs Host Disease | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This is a phase 2, double-blind, randomized (1:1 ratio) study
Who Masked: Participant, Care Provider
Masking Description: Double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adult and pediatric patients who received an allogeneic stem cell transplant (allo-HCT) (Active Comparator): Participants are Allo-HCT recipients
  Interventions: Device: Photobiomodulation Therapy
- Adult and pediatric patients who received a placebo treatment (Placebo Comparator): Participants are Allo-HCT recipients
  Interventions: Other: Placebo sham device

INTERVENTIONS:
Device: Photobiomodulation Therapy — Participants with a history of allo-HCT and diagnosis with oral chronic GvHD randomized to the treatment arm will be treated with oral photobiomodulation/PBM (via Thor LX2.3 system device) for 28 days
  Other Names: PBM Therapy; Thor LX2.3 system device
  Arms: Adult and pediatric patients who received an allogeneic stem cell transplant (allo-HCT)
Other: Placebo sham device — Participants with a history of allo-HCT and diagnosis with oral chronic GvHD randomized to the placebo arm will be treated with a placebo sham device (via Thor LX2.3 sham device setting) for 28 days
  Other Names: Thor LX2.3 sham device setting
  Arms: Adult and pediatric patients who received a placebo treatment

SUMMARY:
The purpose of this study is to find out whether photobiomodulation/PBM therapy using the Thor LX2.3 therapy system is a safe and effective treatment for oral Graft-Versus-Host Disease/GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Allo-HCT recipients
* Age ≥ 4 years-old
* Oral cGvHD with NIH-modified OMRS score ≥ 3 who have failed ≥ 1 line of therapy, including topical corticosteroids..
* No change in systemic immunosuppressive therapy (type or intensity level) within 2 weeks prior to enrollment.
* If a patient is currently using another oral topical treatment for mouth lesions/symptoms, patient must be stable on this treatment for ≥2 weeks prior to study enrollment. Patient may continue same topical dose/frequency during the study period.

Exclusion Criteria:

* Presence of an active uncontrolled infection. Subjects with a controlled infection receiving definitive therapy for 48 hours prior to enrollment are eligible.
* Personal history of mucosal head and neck cancer in the past 5 years.
* Pregnant or breastfeeding.
* The subject or guardian is unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up, and research tests.
* Any serious medical or psychiatric illness that could, in the Investigator's opinion, potentially interfere with the completion of treatment according to this protocol.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Response rate of participants | 28 days
  To assess the primary objective, we will compare the treatment response rates, defined as the the proportion of oral GvHD allo-HCT patients who achieve a CR or a PR at Day 28, for the PBM and Placebo arms. The treatment response rate will be calculated within each study arm for all patients who completed at least one PBM or placebo treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alina Markova, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - National Institute of Health (Data Collection AND Specimen Analysis), Bethesda, Maryland
  - Memorial Sloan Kettering at Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Cancer Center @ Nassau (Consent only), Uniondale, New York
  - University of Pittsburgh Medical Center (Data Collection Only), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
• Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org